CLINICAL TRIAL: NCT06305845
Title: Crowns Fabricated Digitally by CAD-CAM Technology Versus Prefabricated Crowns on Primary Teeth
Brief Title: Digital Crowns Versus Prefabricated Crowns on Primary Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 152012023
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-03

CONDITIONS: Dental Caries in Children
Keywords: digital crowns; zirconia crowns; primary teeth

STUDY DESIGN:
Intervention Model Description: a randomized clinical trial with two parallel arms
Who Masked: Participant
Masking Description: participants will not be informed of which crown they will receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital crowns (Experimental): Crowns that are fabricated digitally by mean of CAD-CAM technology will be placed after preparation.
  Tooth preparation will include 1.5-2 mm. occlusal reduction and proximal contacts will be opened and the entire clinical crown structure will be reduced by 0.8-1.0 mm.and the preparation will be finished with a subgingival finish line.
  Upper and lower arches will be scanned with an intra oral scanner. A third scan of the occlusal bite is then performed in order to establish the patient's occlusion.
  Brilliant Crios composite blocks will be milled with the CEREC MC X milling unit and the inner surface of the crown will be sandblasted followed by etching with 5% hydrofluoric acid for 60 seconds.
  Interventions: Procedure: Digital crowns
- Zirconia crowns (Active Comparator): Prefabricated zirconia crowns that are ready made and supplied in kits with their try-ins will be used in this arm.
  Occlusal reduction of 1.5-2 mm. will be performed by a football diamond bur. The whole crown will be reduced by 0.8-1.0 mm by means of a tapered diamond stone. A shoulder finish line will be created. The try in crown will be tested. Then the shoulder finish line will be removed and the preparation will be extended subgingivally to a feather-edge.
  Interventions: Procedure: zirconia crowns

INTERVENTIONS:
Procedure: Digital crowns — crowns fabricated digitally by CAD-CAM technology
  Other Names: CAD-CAM fabricated crowns
  Arms: Digital crowns
Procedure: zirconia crowns — crowns that are ready made for primary teeth
  Other Names: prefabricated crowns
  Arms: Zirconia crowns

SUMMARY:
Badly decayed primary molars will be treated by performing the pulp therapy technique indicated, then the patients will be randomized into two groups to receive the restorative intervention. For the intervention group, teeth will be prepared to receive the digital crown after intraoral scanning while for the control group, teeth will be prepared to receive the prefabricated zirconia crowns. Teeth will be followed up clinically for 1 year, at 1, 6 and 12 months.

DETAILED DESCRIPTION:
This is a 12-month randomized, controlled, two parallel arms clinical trial. Patients aging from 4 to 10 years with multi-surface decay will be selected. After caries removal and pulp exposure, pulpotomy or partial pulpectomy technique will be performed,then the teeth will be randomized to the interventional group of digital crowns or to the control group of prefabricated zirconia crowns. For preparation of digital crowns, the occlusal reduction was done by 1.5-2 mm. The proximal contacts will be broken and the entire clinical crown structure was reduced by 0.8-1.0 mm , followed by a a subgingival finish line . For the scanning procedure, the upper and lower arches will be scanned with intra oral scanner, and making sure every point is well detailed . A third scan of the occlusal bite is then performed in order to establish the patient's occlusion.

For the milling procedure, Brilliant Crios composite the blocks will be used and milled with the CEREC MC X milling unit . The inner surface of the crown will be sandblasted with Al2O3 .

For zirconia crown preparation, occlusal reduction of 1.5-2mm will be performed by a football diamond bur. The occlusal third of the buccal and lingual surfaces will be also reduced . The whole crown will be reduced by 0.8-1.0 mm by means of a tapered diamond stone .A shoulder finish line will be created. The try in crown will be tested, then the shoulder finish line will be removed and the preparation will be extended subgingivally to feather-edge.

The crowns will then be cemented with the self-adhesive resin cement (Solocem, Coltene, Whaledent, Altstatten, Switzerland) .Light curing was performed while applying pressure on the crown and then waiting for 5 minutes for complete cementing

ELIGIBILITY:
Inclusion Criteria:

* Patients within the age group of 4-10years. Badly decayed or multi-surface affected primary teeth Healthy children free of any systemic disease Patients with cooperative behavior rating definitely positive or positive on the Frank rating scale

Exclusion Criteria:

* Teeth with developmental disturbances
* Teeth with poor prognosis as signs of necrosis, extensive pathological root resorption
* patients with parafunctional habits

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Patient and parent satisfaction | 1, 6 and 12 months
  5-point Likert scale for patient and parent satisfaction.(1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied)

SECONDARY OUTCOMES:
Retention of the crowns | 1, 6 and 12 months
  It will be recorded by clinical examination as a binary outcome; Yes: if crown is retentive & No: if crown is unretentive
Gingival inflammation | 1, 6 and 12 months
  It was measured by gently inserting the tip of a periodontal probe into the sulcus surrounding each crowned tooth. Scoring as follows:
  0 = Normal (Absence of inflammation)
  1. = Mild gingivitis (slight change in color, slight edema. No bleeding on probing)
  2. = Moderate gingivitis (redness, edema and glazing. Bleeding on probing)
  3. = Severe gingivitis (marked redness and edema; ulceration;tendency to spontaneous bleeding
Color match | 1, 6 and 12 months
  The color match will be recorded in natural light with the patient in the upright position for 5 to 10 seconds. No noticeable difference from adjacent teeth, Slight shade mismatch , Obvious shade mismatch and will be recorded digitally by vita easy shade
Opposing tooth wear | 1, 6 and 12 month
  The wear of opposing teeth for the crowns placed will be measured by Smith and Knight Index and it will be measured digitally by a software

CONTACTS AND LOCATIONS:
Overall Officials: Hend Hafez, Professor, Study Director — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
All required data will be published in the manuscript or upon request

REFERENCES:
- [Background] Prabhu D, Anantharaj A, Praveen P, Rani SP, Sudhir R. A clinical and radiographic comparative evaluation of custom-made zirconia crowns using CAD-CAM and stainless steel crowns in primary molars. J Indian Soc Pedod Prev Dent. 2022 Jan-Mar;40(1):34-42. doi: 10.4103/jisppd.jisppd_269_21. PMID 35439881
- [Background] Holsinger DM, Wells MH, Scarbecz M, Donaldson M. Clinical Evaluation and Parental Satisfaction with Pediatric Zirconia Anterior Crowns. Pediatr Dent. 2016;38(3):192-7. PMID 27306242
- [Background] Mourouzis P, Arhakis A, Tolidis K. Computer-aided Design and Manufacturing Crown on Primary Molars: An Innovative Case Report. Int J Clin Pediatr Dent. 2019 Jan-Feb;12(1):76-79. doi: 10.5005/jp-journals-10005-1591. PMID 31496579
- [Background] Al-Halabi MN, Bshara N, Nassar JA, Comisi JC, Rizk CK. Clinical Performance of Two Types of Primary Molar Indirect Crowns Fabricated by 3D Printer and CAD/CAM for Rehabilitation of Large Carious Primary Molars. Eur J Dent. 2021 Jul;15(3):463-468. doi: 10.1055/s-0040-1721905. Epub 2021 Feb 3. PMID 33535245